CLINICAL TRIAL: NCT02733497
Title: Cardiac Autonomic Changes After Endoscopic Thoracic Sympathectomy For Essential Palmar Hyperhidrosis: Results Of A Prospective, Randomized Study
Brief Title: Cardiac Autonomic Changes After Endoscopic Thoracic Sympathectomy For Essential Palmar Hyperhidrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Alfonso Fiorelli, MD, PhD, University of Campania Luigi Vanvitelli
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1185/2011
Record Dates: First submitted 2016-04-05; First posted 2016-04-11 (Estimated); Last update posted 2016-04-12 (Estimated); Status verified 2016-04

CONDITIONS: Hyperhidrosis
Keywords: sympathectomy, sympathicotomy, heart rate variability,
MeSH Terms: conditions — Hyperhidrosis | interventions — Sympathectomy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sympathectomy Group (Active Comparator): Excision of ganglia at T3 level
  Interventions: Procedure: Sympathectomy
- Sympathicotomy Group (Active Comparator): Resection of sympathetic chain at T3 level
  Interventions: Procedure: Sympathicotomy

INTERVENTIONS:
Procedure: Sympathectomy — Resection of ganglia at T3 level
  Arms: Sympathectomy Group
Procedure: Sympathicotomy — Cutting of symptahetic chain at T3 level without ganglia excision
  Arms: Sympathicotomy Group

SUMMARY:
Essential palmar hyperhidrosis (EPH) is a pathological condition of excessive sweating of the hands due to an unexplained over-activity of the T2 and T3 sympathetic fibers. Endoscopy Thoracoscopic Sympathectomy (ETS) is the treatment of choice in patients with EPH refractory to medical treatment .

The cardiac sympathetic activity is mainly controlled by cervical sympathetic fibers but anatomic studies have showed that "accessory" fibers from the T2 and T3 sympathetic ganglia come to the heart and influence its function.

Heart Rate Variability (HRV) is a simple and non-invasive method based on electrocardiogram to evaluate the sympathovagal balance at the sino-atrial level. Several studies have found that ETS caused a decrease of heart rate (HR), an increase of HR variability (HRV) and a shift of sympathovagal balance toward parasympathetic tone but remains unclear if these changes are associated with the extend of ETS.

Thus, in the present study the investigator performed a prospective analysis of HRV function in patients with EPH undergoing different sympathetic denervations as sympathectomy and sympathicotomy with the hypothesis that cardiac autonomic changes could be associated with the extend of sympathetic resection.

DETAILED DESCRIPTION:
It was an unicenter prospective study performed at Thoracic Surgery Unit of Second University of Naples. Patients with severe EPH were randomly assigned to Sympathectomy or Sympathicotomy Group in 1:1 ratio .

Bilateral ETSs were performed in a one-stage procedure by the same surgeon. General anaesthesia using single-lung ventilation technique was performed and patient was placed in standard lateral thoracotomy position. Immediately after the induction of anaesthesia, a local infiltration with 2% lidocaine and epinephrine was injected at each port 5 minutes before the incision to reduce postoperative pain. The first port was placed in the 3th intercostal space below and anterior to inferior angle of scapula and through that a 10 mm 30 degree camera was inserted. A second 5 mm working port was placed at the same intercostal space in the anterior axillary line. After identification of sympathetic chain, in Sympathectomy Group the T3 ganglion was excised at the top of the third rib while in Sympathicotomy Group the sympathetic chain was resected between T2-T3 ganglia at the same level but the T3 ganglion was left intact. At the end of the procedure, a 16 F drainage was inserted through the port and the lung was re-inflated to allow the air drainage from pleural cavity and to prevent pneumothorax. The drain was subsequently removed.

All measurements on cardiac autonomic function were performed one week before ETS and different post-operative time-points (7 days, 1, 3 and 6 months after ETS). The results were prospectively registered and then retrospectively analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Age more than 18 years
* Severe hyperhidrosis

Exclusion Criteria:

* Contraindications for general anaesthetic procedure and/or for selective endotracheal intubation
* Previous pleural or lung diseases that make difficult the access to pleural cavityù
* Cardiac diseases and/or taking medications with cardiac effects
* Secondary hyperhidrosis including hyperthyroidism, acute and chronic infections, malignancy, and immunologic disorder
* Mild or moderate palmar hyperhidrosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-01; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Heart Rate (HR) measured in beats/min | 7 days, 1, 3 and 6 months after operation

SECONDARY OUTCOMES:
Post-operative complications | Post-operative time and 7 days, 1, 3 and 6 months after operation
Compensatory hyperhidrosis measured with a scale ranging from 0 (absent) to 3 (severe) | 1, 3 and 6 months after operation

CONTACTS AND LOCATIONS:
Overall Officials: Mario Santini, MD, Study Chair — University of Campania Luigi Vanvitelli

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Katara AN, Domino JP, Cheah WK, So JB, Ning C, Lomanto D. Comparing T2 and T2-T3 ablation in thoracoscopic sympathectomy for palmar hyperhidrosis: a randomized control trial. Surg Endosc. 2007 Oct;21(10):1768-71. doi: 10.1007/s00464-007-9241-9. Epub 2007 Apr 3. PMID 17404794
- [Background] Tedoriya T, Sakagami S, Ueyama T, Thompson L, Hetzer R. Influences of bilateral endoscopic transthoracic sympathicotomy on cardiac autonomic nervous activity. Eur J Cardiothorac Surg. 1999 Feb;15(2):194-8. doi: 10.1016/s1010-7940(98)00309-1. PMID 10219553
- [Background] Cruz J, Sousa J, Oliveira AG, Silva-Carvalho L. Effects of endoscopic thoracic sympathectomy for primary hyperhidrosis on cardiac autonomic nervous activity. J Thorac Cardiovasc Surg. 2009 Mar;137(3):664-9. doi: 10.1016/j.jtcvs.2008.07.021. Epub 2008 Sep 24. PMID 19258086
- [Derived] Fiorelli A, Messina G, Chiodini P, Costanzo S, Viggiano A, Monda M, Vicidomini G, Santini M. Cardiac Autonomic Changes After Thoracic Sympathectomy: A Prospective, Randomized Study. Ann Thorac Surg. 2017 Jan;103(1):216-224. doi: 10.1016/j.athoracsur.2016.10.055. Epub 2016 Nov 23. PMID 27889103